CLINICAL TRIAL: NCT01382550
Title: Prevention of Recurrent Venous Thromboembolism in Patients With Low Circulating Levels of Antithrombin. Extended Anticoagulation vs 12-Month Oral Anticoagulation
Brief Title: Prevention of Thrombosis Recurrence in Patients With Low Circulating Levels of Antithrombin.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Giovanni Di Minno, Director of the Dept of Clinical and Experimental Medicine, Federico II University
Other Study IDs: AT 63/11
Record Dates: First submitted 2011-06-23; First posted 2011-06-27 (Estimated); Last update posted 2012-09-13 (Estimated); Status verified 2012-09

CONDITIONS: Venous Thrombosis
Keywords: antithrombin; venous thrombosis; thrombosis risk factors; thrombophilia
MeSH Terms: conditions — Venous Thrombosis; Thrombophilia | interventions — Ornithine-Oxo-Acid Transaminase

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- VTE subjects: subjects with a recent (<3 months) first VTE event undergoing long-lasting OAT or 12-month OAT
  Exclusion criteria: missing data during the follow-up; contraindications to or lack of compliance to oral anticoagulation (OAT), lack of informed consent; history of previous VTE event; indication for continuous oral anticoagulation (e.g., an artificial heart valve or chronic atrial fibrillation); events occurring during pregnancy, malignancy, puerperium, oral contraceptive intake, hormone replacement therapy; deficiencies of Prot. C and Prot S or combined inhibitor deficiencies.
  Interventions: Drug: long-lasting OAT or 12-month OAT

INTERVENTIONS:
Drug: long-lasting OAT or 12-month OAT — The antithrombotic treatment will be decided according to usual practice of enrolling Centers. The duration of the initial treatment with parenteral anticoagulation (Low Molecular Weight Heparin or Fondaparinux), the beginning of oral anticoagulation (OAT) with Vit K inhibitors and the International Normalized Ratio (PT-INR) target will be recorded.
  According to Center indications the OAT duration (6 months, 12 months or long-lasting) will be recorded and population will be stratified accordingly. The length of therapy will be counted from the date when a stable PT-INR is achieved.
  The occurrence of surgery, trauma, prolonged immobilization (>7 days), pregnancy (VTE risk periods) during the follow-up and the use of adequate anti-thrombotic prophylaxis will be recorded.

SUMMARY:
The aim of this study is to estimate the incidence of spontaneous and provoked recurrent VTE and the bleeding events during a 10-year follow-up in subjects experiencing a first VTE stratified according to % AT levels and to treatment schedule (long-term vs 6-12 months oral anticoagulation+transient prophylaxis during high risk periods)

DETAILED DESCRIPTION:
Study population: subjects with a recent (<3 months) first VTE event will be enrolled for a long-term follow-up. Clinical visits will be performed every 4-6 months (average).

In each case, objective diagnosis has to be achieved by compression ultrasonography, the diagnosis being based on the lack of compressibility of one or more venous segments. PE has to be documented by ventilation/perfusion lung scanning or by spiral computed tomography (CT).

For each subject, information about pregnancy, active malignancy, recent (<3 mo) surgery or trauma, fracture, immobilization, acute medical illness, use of oral contraceptives, long-distance travel, personal or family history of arterial and/or venous thrombosis or repeated birth losses will be collected. In the presence of at least one of the previous risk factors, VTE will be defined as secondary otherwise idiopathic. Further information, collected from the whole population by a trained staff, were the following: gender, age, weight, height, body mass index (BMI), waist circumference, personal history of symptomatic atherosclerosis (i.e. ischemic stroke, transient ischemic attack, acute myocardial infarction, angina, intermittent claudication), arterial hypertension, use of antihypertensive drugs, diabetes mellitus, use of antidiabetic drugs, hyperlipidemia, use of statins, smoking habit (use of cigarettes/d), current use of heparin, use of oral anticoagulant (how long) or of antiplatelet drugs (how long), chronic consumption of other drugs.

All these information will be collected by a trained staff on admission and during follow-up visits (every 4-6 months).

Exclusion criteria: missing data during the follow-up; contraindications to or lack of compliance to oral anticoagulation (OAT), lack of informed consent; history of previous VTE event; indication for continuous oral anticoagulation (e.g., an artificial heart valve or chronic atrial fibrillation); events occurring during pregnancy, malignancy, puerperium, oral contraceptive intake, hormone replacement therapy; deficiencies of Prot. C and Prot S or combined inhibitor deficiencies.

Laboratory Studies All laboratory evaluations will be carried out at least 2 weeks after cessation of the anticoagulant therapy or after a switching to low-molecular weight heparin (LMWH) treatment. Antithrombin (AT) functional activity will be measured and VTE patients will be stratified into 3 subgroups of AT% (1st: <70%, 2nd: 70-80, 3rd: >81%). AT measurements will be confirmed in a second sample collected 3 months later. In case of discrepancy between the results of the 2 tests, a third sample will be collected. Protein C and S; antiphospholipid antibodies (IgG and IgM); homocysteine, and factor V Leiden and prothrombin 20210A polymorphisms will be determined using commercially available kits by technicians who had been unaware of the patients' treatment assignments and of the clinical course.

Antithrombotic treatment The antithrombotic treatment will be decided according to the usual practice of the enrolling Center. The duration of the initial treatment with parenteral anticoagulation (Low Molecular Weight Heparin or Fondaparinux), the beginning of oral anticoagulation (OAT) with Vit K inhibitors and the International Normalized Ratio (INR) target will be recorded.

According to Center indications the OAT duration (6 months, 12 months or long-lasting) will be recorded and population will be stratified accordingly. The length of therapy will be counted from the date when a stable prothrombin time within the target INR range is achieved.

The occurrence of surgery, trauma, prolonged immobilization (>7 days), pregnancy (VTE risk periods) during the follow-up and the use of adequate anti-thrombotic prophylaxis will be recorded.

Follow-up Subjects will be followed-up at 3, 6, and 12 months after enrollment and at least every 6 months thereafter either by a visit to the Center or by telephone contact. INR values will be reported by telephone twice monthly. At each visit the patients will be asked about new symptoms of VTE and about bleeding manifestations. When appropriate, a clinical assessment will be made and diagnostic tests will be performed.

Information on major and minor bleedings during oral anticoagulation will be collected in the whole sample. Major bleedings will be defined as hemorrhages that were either retroperitoneal or intracranial or associated with a decrease in hemoglobin of at least 2.0 g per deciliter or that had required either transfusion of at least 2 units of blood (or of red cells) or an invasive procedure, including surgery, to stop them or if they warranted permanent OAT withdrawing.

Study end points The incidence of objectively documented recurrent VTE (DVT and/or PE) during the life-long follow-up is the primary outcome of this study. Contralateral DVT and PE will be computed as a recurrence. Ipsilateral DVT will be adjudicated recurrent if the results of the tests are worse than those obtained in a previous test or if the thrombus is diagnosed in another venous district of the leg. DVT of the arm; CT or MRI-documented occlusion of cerebral/abdominal veins; ultrasound-documented thrombosis of the great saphenous vein of the leg not involved in the first appearance will be also defined as a recurrence. The total (minor and major) bleeding occurrence during the life-long follow-up represents the safety end-point of this study and will be analyzed according to the thrombolysis in myocardial infarction (TIMI) bleeding score.

Sample size Assuming a 20:1:1 sample size ratio between AT% subgroups (AT%> 80%; AT%=70-80%; and AT%<70%, respectively), to detect an increase in the incidence of recurrent events from 0.3 in the control population (AT% > 80%) to 0.6 in each of the other two subgroups (AT%=70-80% and AT%<70%), a sample size of about 900 subjects is needed (power= 95%; α=0.025, to allow for two independent comparisons).

Expected results Among individuals with a history of first VTE stratified according to AT% levels, the risk/benefit analysis of this study will help identify group(s) of individuals with a strong indication to long-term oral anticoagulation.

ELIGIBILITY:
Inclusion Criteria:

* Recent (<3 months) First VTE event

Exclusion Criteria:

* missing data during the follow-up; contraindications to or lack of compliance to oral anticoagulation (OAT), lack of informed consent; history of previous VTE event; indication for continuous oral anticoagulation (e.g., an artificial heart valve or chronic atrial fibrillation); events occurring during pregnancy, malignancy, puerperium, oral contraceptive intake, hormone replacement therapy; deficiencies of Prot. C and Prot S or combined inhibitor deficiencies.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: subjects with a recent (<3 months) first VTE event enrolled for a long-term follow-up (every 6 months).
Sampling Method: Non-Probability Sample
Enrollment: 900 (Estimated)
Dates: Start 1993-03; Primary Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
VTE recurrence during the 8-year follow-up | At an average of 8 years of follow-up
  During the 8-years follow-up, the incidence of recurrent VTE will be evaluated stratifying population according to OAT treatment and AT%. Contralateral DVT and PE will be computed as a recurrence. Ipsilateral DVT will be adjudicated recurrent if the results of the tests are worse than those obtained in previous tests or if the thrombus is diagnosed in another venous district. DVT of the arm; CT or MRI-documented occlusion of cerebral/abdominal veins; ultrasound-documented thrombosis of the great saphenous vein of the leg not involved in the first appearance will be also defined as a recurrence

SECONDARY OUTCOMES:
Bleeding events during the 8-year follow-up | During the 8-year follow-up
  During the 8-years follow-up, the incidence of overall (minor and major) bleedings will be evaluated stratifying population according to OAT treatment and AT%. The severity of bleeding events will be defined according to the thrombolysis in myocardial infarction (TIMI) bleeding score.

CONTACTS AND LOCATIONS:
Overall Officials: Giovanni Di Minno, Prof, Study Chair — Federico II University; Matteo Nicola Dario Di Minno, MD, Principal Investigator — Federico II University; Anna Maria Cerbone, MD, Principal Investigator — Federico II University; Antonella Tufano, MD, Principal Investigator — Federico II University
Locations (1):
- Federico II University, Naples, Italy, Italy

REFERENCES:
- [Derived] Di Minno MN, Dentali F, Lupoli R, Ageno W. Mild antithrombin deficiency and risk of recurrent venous thromboembolism: a prospective cohort study. Circulation. 2014 Jan 28;129(4):497-503. doi: 10.1161/CIRCULATIONAHA.113.003756. Epub 2013 Oct 21. PMID 24146249